CLINICAL TRIAL: NCT04848779
Title: A Prospective Observational Study to Describe Clinical Outcomes of Alglucosidase Alfa Treatment in Patients ≤6 Months of Age With Infantile-onset Pompe Disease (IOPD)
Brief Title: A Prospective Study to Observe & Describe Clinical Outcomes of Alglucosidase Alfa Treatment in Patients ≤6 Months of Age With Infantile-onset Pompe Disease (IOPD)
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17003; U1111-1266-4848 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-03-29; First posted 2021-04-19 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Glycogen Storage Disease Type II
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 104 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1
  Interventions: Drug: Alglucosidase alfa GZ419829

INTERVENTIONS:
Drug: Alglucosidase alfa GZ419829 — Pharmaceutical form: Lyophilized powder for solution
  Route of administration: intravenous
  Other Names: Myozyme

SUMMARY:
Primary Objective:

To describe the effect of routine practice with alglucosidase alfa in patients with IOPD ≤6 months of age, on invasive ventilation-free survival after 52 weeks of treatment.

Secondary Objectives:

* To describe the effect of routine practice with alglucosidase alfa on invasive ventilation-free survival and survival at 12 and 18 months of age, as well as on change in left ventricular mass (LVM) Z score, Alberta Infant Motor Scale (AIMS) score, body weight, body length, and head circumference Z scores, and urinary glucose tetrasaccharide (Hex4), at Week 52 of treatment.
* To describe the safety, tolerability, and immunogenicity of alglucosidase alfa in the routine practice of IOPD treatment.

DETAILED DESCRIPTION:
The planned duration of observation for each participant will be 104 weeks after enrollment, to determine secondary outcomes at 18 months (approximately 78 weeks) of age.

ELIGIBILITY:
Inclusion Criteria:

* At the time of informed consent, participants must be ≤6 months of age, corrected for gestation if necessary. Gestational age <40 weeks will be adjusted to a full-term gestational age of 40 weeks.
* Participants must have alglucosidase alfa enzyme replacement therapy (ERT) planned or initiated for IOPD treatment irrespective of study participation, according to the treating physician's decision regarding participants' routine disease management.
* Participants must have available and accessible medical records from the time of IOPD diagnosis and from subsequent follow-up.
* Participants must have a confirmed diagnosis of IOPD, defined as presence of 2 pathogenic acid alpha glucosidase (GAA) variants and documented GAA deficiency in blood (dried blood spot [DBS] accepted), skin, or muscle tissue, or presence of 1 pathogenic GAA variant and documented GAA deficiency in blood, skin, or muscle tissue from separate samples (either from 2 different tissues or from the same tissue but at 2 different sampling dates.) (DBS and leukocytes are acceptable as 2 different samples from blood).
* Participants must have established cross-reacting immunologic material (CRIM) status available prior to enrollment. CRIM status may be provided by historical CRIM testing results or prediction of CRIM status based on genotyping performed at a Clinical Laboratory Improvement Amendments (CLIA) or other appropriately certified genetic laboratory.
* Participants must have cardiomyopathy at the time of diagnosis (LVMI equivalent to mean age-specific LVMI):

  * LVMI +1 standard deviation (SD) in participants diagnosed by newborn or sibling screening,
  * LVMI +2 SD in participants diagnosed by clinical evaluation.
* Participants must have informed consent provided by parent(s)/legally acceptable representatives (LARs).

Exclusion Criteria:

* Participants with respiratory insufficiency, defined as:

  * Oxygen saturation <90% on room air as determined by pulse oximetry,
  * Venous partial pressure of carbon dioxide (pCO2) >55 mmHg or arterial pCO2 >40 mmHg on room air,
  * Use of invasive (with intubation or tracheostomy) or noninvasive (no intubation or tracheostomy) ventilation at enrollment, for participants not having started ERT at enrollment,
  * Use of invasive or noninvasive ventilation at the time of ERT initiation, for participants having started ERT before enrollment.
* Participants with major congenital abnormality including heart defect, neural tube defect, or Down syndrome that, in the opinion of the investigator, would preclude participation in the study or potentially decrease survival.
* Participants with clinically significant organic disease other than signs/symptoms related to Pompe disease, including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or circumstance that, in the opinion of the investigator, would preclude participation or potentially decrease survival.
* Previous or ongoing treatment in any clinical trial of, or managed access program for, avalglucosidase alfa or any other Pompe disease-specific therapy.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 0 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Confirmly diagnosed IOPD patients 6 months or less of age (corrected for gestational age if needed), treated or planned to be treated with alglucosidase alfa, at the time of study inclusion.
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2026-10-28 (Estimated); Study Completion 2026-10-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants alive and free of invasive ventilation at Week 52 of treatment | Week 52

SECONDARY OUTCOMES:
Proportion of participants alive and free of invasive ventilation at 12 and 18 months of age | at 12 and 18 months of age
Proportion of participants alive at Week 52 of treatment | Week 52
Proportion of participants alive at 12 months and 18 months of age | at 12 and 18 months of age
Proportion of participants free of ventilator use and free of supplemental oxygen use at Week 52 | Week 52
Change from baseline to Week 52 in LVM Z score | from baseline to Week 52
Change from baseline to Week 52 in AIMS score | from baseline to Week 52
Change from baseline to Week 52 in body length Z-scores | from baseline to Week 52
Change from baseline to Week 52 in body weight Z-scores | from baseline to Week 52
Change from baseline to Week 52 in head circumference Z-scores | from baseline to Week 52
Change from baseline to Week 52 in body length percentiles | from baseline to Week 52
Change from baseline to Week 52 in body weight percentiles | from baseline to Week 52
Change from baseline to Week 52 in head circumference percentiles | from baseline to Week 52
Change from baseline to Week 52 in urinary Hex4 | from baseline to Week 52
Number of participants experiencing at least 1 treatment-emergent adverse events (TEAE), including infusion-associated reactions (IAR) | From inclusion for 104 weeks
Number of participants with abnormalities in physical examinations | From inclusion for 104 weeks
Number of participants with abnormalities in clinical laboratory results | From inclusion for 104 weeks
Number of participants with abnormalities in vital signs measurements | From inclusion for 104 weeks
Number of participants with abnormalities in 12-lead electrocardiogram (ECG) | From inclusion for 104 weeks
Incidence of treatment-emergent antidrug antibodies (ADA) | From inclusion for 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- United States (5):
  - Advanced Medical Genetics- Site Number : 8400002, Hawthorne, New York
  - Duke University Medical Center- Site Number : 8400004, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center- Site Number : 8400001, Cincinnati, Ohio
  - Le Bonheur Children's Hospital- Site Number : 8400005, Memphis, Tennessee
  - Seattle Children's Hospital- Site Number : 8400003, Seattle, Washington
- Investigational Site Number : 0560001, Leuven, Belgium
- Investigational Site Number : 2500001, Tours, France
- Investigational Site Number : 2760001, Giessen, Germany
- Italy (2):
  - Investigational Site Number : 3800002, Monza, Monza E Brianza
  - Investigational Site Number : 3800001, Florence
- Investigational Site Number : 5280001, Rotterdam, Netherlands
- Investigational Site Number : 7240001, Esplugues de Llobregat, Catalunya [Cataluña], Spain
- Investigational Site Number : 1580001, Taipei, Taiwan
- United Kingdom (2):
  - Investigational Site Number : 8260001, London, London, City of
  - Investigational Site Number : 8260002, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org